CLINICAL TRIAL: NCT02214511
Title: Etude de la sensibilité Aux Signaux Sociaux Dans la dépression, Modulateurs Psychologiques, Comportementaux et Inflammatoires.
Brief Title: Biomarkers of Social Sensitivity in Major Depression
Acronym: SENSO
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C13-31; 2013-A01484-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2014-06-30; First posted 2014-08-12 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; social rejection; rapid facial reaction; facial mimicry; prosocial behavior; inflammation; self esteem
MeSH Terms: conditions — Depressive Disorder, Major; Social Isolation; Altruism; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to explore inflammatory cytokines. Dosage of IL-6, IL-10, TNFa, IP-10, MCP-1, MIP-1b, Rantes, sIL-6Ra, IL1ra, VEGF, Leptin, PECAM1, sTie2, sVEGFR1, sVEGFR2 will be performed by luminex technique and usCRP, srIL2 ans sCD14 by ELISA technique.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MDD patients: emotional facial stimuli cyberball game
  Interventions: Behavioral: emotional facial stimuli; Behavioral: Cyberball game
- healthy subjects: emotional facial stimuli cyberball game
  Interventions: Behavioral: emotional facial stimuli; Behavioral: Cyberball game

INTERVENTIONS:
Behavioral: emotional facial stimuli — Subjects watch passively dynamic facial emotions obtained by emotionnal faces photos morphing. Their rapid facial reactions are recorded by faciel EMG device as eye movement by occulometric device.
Behavioral: Cyberball game — Ball tossing computer game to manipulate social inclusion status : rejection or inclusion. Social behavior, social pain and inflammatory modification will be assessed after the game.

SUMMARY:
Major depression disorder (MDD) is a frequent and disabling mental disorder with great risk of recurrence and chronicity. Interpersonal factors are among the strongest predictors of the course and duration of an episode of depression. More specifically, social rejection is one of the most environmental risk factors of MDD. Targeted rejection predicts hastened onset of major depression. On the other hand, healthy subject show prosocial behavior after social rejection to reconnect to new source of social interaction. In addition to the potential impact of social exclusion on MDD onset, depressed patients may be more prone to be rejected as they encounter interpersonal difficulties and may less be able to reconnect to the social group after rejection.

Recent neuroimaging data show that brain processing of social exclusion activate brain regions that are central to the pathophysiology of MDD. Some of these regions are also known to be activated during physical pain and may contribute to the aversive dimension of the experienced rejection. Pro-inflammatory cytokines are involved in MDD physiopathology and can induce social withdrawal behavior. Inflammation can modulate social interactions in mammals. Moreover, after a social stress such as social rejection, blood cytokines increase. At a cognitive level, self-esteem can modulate the sensitivity to social rejection.

The major objective of the trial is to study sensitivity to social signals in MDD patient compared to healthy subject.

The investigators hypothesize in MDD patient : (1) decrease of rapid facial reactions (RFR) to dynamic emotional faces expressing joy, (2) increase of RFR to dynamic emotional faces expressing sadness, (3) decrease of prosocial reaction after experimental social rejection.

Secondary objective is to identify psychological and biological mediators We hypothetize in MDD patient: (1)mediating effect of systemic inflammatory cytokines, an (2) mediating effect of state self esteem 30 MDD patients and 60 healthy subject will be included. They will encounter psychiatric and psychometric evaluation. Their facial EMG will be recorded to assess RFR to dynamic emotional faces created by photo morphing from KDEF emotional faces database, coupled to occulometric recording. Subjects will perform cyberball game as an experimental inclusion or exclusion task and the trustgame task as an implicit evaluation of their prosocial behavior. Questionnaires will assess explicit measurement of social rejection pain and desire of affiliation. Inflammatory markers will be measured in a blood sample before the cyberball task for every subjects and 6 hours later for 20 healthy volunteers. Dosage of IL-6, IL-10, TNFa, IP-10, MCP-1, MIP-1b, Rantes, sIL-6Ra, IL1ra, VEGF, Leptin, PECAM1, sTie2, sVEGFR1, sVEGFR2 will be performed by luminex technique and usCRP, srIL2 ans sCD14 by ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

For everybody :

* benefit social health insurance
* french speaker and reader
* can stop smoking one day
* volunteer to participate

For 1st group :

* actual MDD diagnosed by a psychiatrist and meet the DSM IV criterias of MDD
* no antidepressant treatment or antidepressant treatment for less than 7 days.

Exclusion Criteria:

* BMI > 40
* weekly sport > 3 hours
* pregnancy
* fever or other infection symptoms during the last month
* significant or unstable disease, especially neurologic or inflammatory.
* recent history of coronary disease, ulcer, COPD, severe dyslipemia, kidney or liver failure.
* severe smoking addiction (fagerström > 8)
* antiinflammatory or immunomodulatory treatment during last month

For 1st group :

* no psychiatric treatment except benzodiazepin if no severe vigilance trouble and antidepressant treatment more than 7 days
* subjects under legal protection
* constraint hospitalization
* significant suicidal risk
* resistant MDD
* psychiatric comorbidity

For 2nd group :

- psychiatric disease, actual or past according to DSM IV criterias

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. st group : major depression disorder patients
  2. nd group : healthy volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Rapid facial reactions : milliVolts amplitude of electromyographic signal of zygomaticus, corrugator, depressor & frontalis muscles | During stimuli presentation (emotional faces) at Day 1 from 9:40 to 10:30 am
  During passive watching of dynamic emotional faces, electromyographic signal is recorded with skin electrodes facing zygomaticus, corrugator, depressor & frontalis muscles.
Implicit pro-social behavior : invested money during a 4-round trust game | At Day 1 from 11:40 to 11:50 am
  Total amount of money invested by the subject during a 4-round trust game without feedback.
Explicit pro-social behavior : affiliation desire measured by a questionnaire | At Day 1 from 11:50 to 12:00 am
  Affiliation desire questionnaire from Park and Manner assessing total affiliation desire and affiliation desire towards close relationship or strangers.

SECONDARY OUTCOMES:
Self esteem assessed by questionnaires mediates social pain after rejection and pro-social behavior | 2 assessments at Day 1 : at 8:30 and at 11:50 am
  Scoring of questionnaires of state and trait self esteem (state self esteem scale and Rosenberg scale)
Systemic inflammation mediates social pain after rejection and pro-social behavior | At day 1 : at 11:30 am and 5:30 pm
  Inflammatory dosage in blood :
  * IL-6, IL-10, TNFa, IP-10, MCP-1, MIP-1b, Rantes, sIL-6Ra, IL1ra, VEGF, Leptin, PECAM1, sTie2, sVEGFR1, sVEGFR2 by luminex technique
  * usCRP, srIL2 ans sCD14 by ELISA technique.

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Pitié Salpêtrière Hospital, Paris, France